CLINICAL TRIAL: NCT03570372
Title: Internet-based Treatment for Adults With Autism Spectrum Disorder (MILAS)
Brief Title: Internet-based Treatment for Adults With Autism Spectrum Disorder.
Acronym: MILAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: Örebro University, Sweden (Other); Regional Research Council Mid Sweden (Unknown); Fredrik och Ingrid Thurings Stiftelse (Unknown); Stiftelsen Professor Bror Gadelius Minnesfond (Unknown)
Responsible Party: Principal Investigator, Fredrik Holländare, Doctor of Philosophy, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17RS4920
Record Dates: First submitted 2018-01-29; First posted 2018-06-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Life quality; ASD; Internet based treatment; Autism; ICBT
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 18 week internet-based CBT with therapist support. Regular online group discussions.
  Interventions: Behavioral: Internet-based treatment for adults with autism spectrum
- Control group (Active Comparator): Reads 2 books about Autism Spectrum Disorder (ASD)
  Interventions: Behavioral: Psychoeducation about autism spectum disorder

INTERVENTIONS:
Behavioral: Internet-based treatment for adults with autism spectrum — Internet-based CBT. The intervention includes 18 modules focusing on: Psychoeducation, individual goal setting, behavioral change, management strategies and stress management
  Arms: Intervention group
Behavioral: Psychoeducation about autism spectum disorder — Self-studies by reading the book "What does the disability mean ?: Living with autism / Asperger syndrome. Project Empowerment "(2004), by Norrö & Swing Åström, as well as a book of biographical stories of people who have ASD. The first book will be read during the first half of the project, and the second will be in the second half.
  Arms: Control group

SUMMARY:
The group of patients diagnosed with Autism spectrum disorder (ASD) is increasing and so is the need for new and effective treatment methods. ASD is characterized, among other things, by difficulties in social interaction and communication. These difficulties often affects their quality of life and causes a risk of developing social anxiety or other forms of mental illness, which often leads to isolation and may cause difficulties in participating in regular face- to- face psychological treatment. Although research shows that group therapy is favorable for this group of patients, many with ASD refrain from group-treatment due to social anxiety or difficulties with public transport. In order to increase the availability of evidence based psychological treatment for these patients, it seems important to be able to offer a web-based treatment option, with the ability to participate in online group sessions.

The aim of the study is to investigate whether Internet-based CBT is an effective method of improving the quality of life and sense of coherence and decreasing symtoms of anxiety and depression among adults with ASD.

A randomized controlled study design will be used. Assessment will be conducted through video interviews, recruiting 84 patients with ASD and normal intellectual abilities. Symptoms of depression and other forms of psychopathology will be assessed through MINI-7 interviews. Primary outcome measures are quality of life. Participants in the intervention group receives a 18 week blended treatment combining individual ICBT delivered through a treatment platform called Stöd och Behandling (SOB) with the opportunity to participate in regular group discussions delivered through a discussion forum online. Participants in the control groups are offered self-studies through psycho educative books about ASD. Data will be collected at baseline, mid-treatment, post-treatment and after six and 12 months.

DETAILED DESCRIPTION:
Background Autism Spectrum Disorder (ASD) is characterized by significant difficulties in social interaction and communication as well as routine boundaries and constraints in behavioral patterns. People with ASD have difficulties in the ability to mentalize, i.e. difficulties in understanding how another person feels and thinks. Another characteristic of persons with ASD is that they are detailed in their way of processing information and therefore have difficulties in generalizing and managing changes in everyday life. Lacking in planning, organizing, evaluating and adjusting their behaviors can lead to extensive needs of support. About 40% of adult patients with ASD exhibit depressive symptoms, and different types of anxiety disorders are also very common. Many people experience constant stress and vigilance following efforts to behave socially adequately and managing unpredictable situations. The difficultiess is often combined with chronic stress and experience of failures and misunderstandings. In addition to having difficulties in socializing, many also have difficulties in initiating and solving problems, which contributes to unemployment.

Psychological treatment Many people with ASD find it difficult to identify and express feelings and thoughts, which is a common element in psychotherapeutic treatment. This can hinder psychological treatment from progressing as expected. The goals of treatment are often to increase the person's quality of life and ability to live an independent life, and a major focus in treatment for children with ASD is on psycho education, cognitive interventions and social skills. Treatment of adults with ASD is less explored. Experience from clinical practice suggests that psychological interventions should be practical and focused on behavioral change strategies, but to date, few treatments using Cognitive Behavioral Therapy (CBT) have been scientifically evaluated for persons with ASD.

A group format has been considered to have several benefits in psychological treatment for adults with ASD. It offers an opportunity for participants to discover that they are not alone in their quest to fit in socially. A group also provides the opportunity to reproduce problematic social situations, provide behavioral feedback and enable exercises of skills in a structured environment.

In several studies, internet based psychological treatment has proven to be effective in treating a variety of psychiatric diagnoses. Courses and information-based training materials have been offered in some regions in Sweden, but only for children and adolescents with ASD. Until now, no internet based cognitive behavioral treatment (ICBT) has been used for treating adults with ASD. Since many with ASD have severe social anxiety or having difficulty with travel, it seems important to be able to offer a web-based treatment option. This could enable social interaction, learning and a sense of belonging, regardless of where they live and the ability to leave the home as well as contributing to a more equal care.

Earlier study A swedish research group have developed a group based CBT manual (called ALMA) for adults with ASD. The treatment aims to give participants a deep understanding of the diagnosis and increase their quality of life. A randomized controlled study of this treatment has been published in a reputable journal . Groups of 6-8 adults with ASD received the intervention for a total of two semesters. The treatment significantly improved the quality of life (Cohen's d = 0.43) and in a cumulative long-term follow-up (> 8 months), it was found that the improvement was lasting. In addition, 88% of the participants gained increased self-understanding, higher self-acceptance (72%) and increased well-being (67%).

Current study

The current study originates from the above-mentioned ALMA treatment. The CBT based material used in ALMA has been transformed and adapted to an internet-based format. The effects of the internet-based version will be evaluated using the same population as in the ALMA study - i.e. adults with ASD.

Purpose The purpose of the study is to investigate whether Internet-based CBT is feasible and effective in improving the quality of life and sense of coherence and decreasing symtoms of anxiety and depression among adults with ASD. Since internet based treatment is relatively unexplored for patients with ASD, we will also investigate the patients' subjective experience of such treatment, as well as systematically investigate what the written communication between patient and therapists will contain.

Research questions

1. Will adults with autism spectrum disorder follow an internet-based individual therapy that includes the possibility of participating in group sessions online for two semesters and, if so, will they experience it as meaningful?
2. Will an internet-based treatment lead to a greater increase in quality of life compared to an active control group, and will this difference remain at follow-up after 6 and 12 months?
3. Will an internet-based treatment lead to decreased symptoms of depression and anxiety compared to an active control group and will this differences remain at follow up?
4. How do participants experience internet-based treatment?
5. What content does the written communication between therapists and participants have?

Method

Design and selection Randomized controlled treatment design with two conditions. The experiment group receives internet-based individual treatment with the possibility of participating in group discussions online. An active control group reads two books about ASD, one describing ASD and the other are stories of individuals who themselves have ASD. 84 persons with ASD between 16 and 55 years will be recruited from all over the country. Exclusion criteria are ongoing psychotherapy with CBT or social behavior training, serious mental illness, mental developmental disorder or high risk of suicide. Additional exclusion criteria include inability to fill out forms and answer questions on the internet and inability to read and understand the Swedish language. Participants will either be randomized into the intervention group or active control group.

Recruitment Information about the project is given to personnel working with the patient group in psychiatric and habilitation centers. Information will also be available in waiting rooms of healthcare facilities, in social media and on websites for psychiatric and autism-related associations, as well as through local press advertising. Potential participants will themselves submit an application of interest to participate via 1177.se, the website for Swedish healthcare e-services. Assessment interviews will be conducted through video link and symptoms of depression and other forms of psychopathology will be assessed through MINI-7 interviews.

Intervention

The intervention group receives 18 modules of internet based CBT (ICBT). The modules and excersices following every module will be provided in text. Each participant has a personal therapist who guides the participant throughout the treatment and provides support and feedback in connection to each completed module of the treatment. The modules contain the following themes:

* Psychoeducation - diagnostic criteria, symptoms, mentalization, perception etc
* Social interaction - relations, communication
* Mental health/illness - depression, anxiety
* Goal settings- individual goals, what can i change?
* Behavioral change - problem solving strategies, functional analyses
* Life style - food, sleep, physical activity
* Stress management - relaxation exercises and energy balancing.
* Everyday strategies - facilitate everyday life, structure and organization
* Social and civil rights - housing support, job opportunities.

The sessions with group discussions will be held at a certain time every 2nd week. The discussions revolve around specific questions linked to the theme of the current treatment week. The discussions will be supervised and led by a therapist and are held through a closed discussion forum online.

Control group The control group is offered self-studies by reading the book "What does the disability mean ?: Living with autism / Asperger syndrome", as well as a book containing biographical stories from people who themselves have ASD. The first book will be read during the first half of the project, and the second will be in the second half.

Power Calculation The experience of treatment for adults with ASD is very limited, and therefore, there are quite few previous results to be based on when making assumptions about the expected effect. However, a previous study of adult patients with ASD found an effect size of d = 0.43 (SD = 1.68) on self-assessed quality of life, measured before and after CBT in group. To get 80% power to find a difference of that size (given an alpha level of 0.05), 42 participants will be recruited. In the previous study (on site) there was a loss of 17%. It is difficult to estimate how much the loss occurs when the treatment is administered through internet, but if assumed that the loss is 50%, the intention is to include at least 84 participants in order to answer the scientific questions. The calculations are made using the PS - Power and Sample Size Calculations software.

Data Collection Each potential participant will initially be asked to answer a questionnaire online. The questionnaire includes questions about psychiatric symptoms, quality of life, demographic variables, employment and knowledge about ASD etc. Information that verifies the ASD diagnosis is obtained from the patients' medical record with the participant's consent. An interview via telephone is conducted with all potential participants and they are interviewed with a structured assessment tool for psychiatric diagnostics (M.I.N.I. version 7). Data on patient satisfaction with treatment and possible side effects are obtained after the end of treatment.

Measurement Quality of life is measured by Brunnsviken Brief quality of Life questionnaire (BBQ) and RAND-36 before and after the end of treatment and in a 6-month and one-year follow-up. EQ-5D and Sense of Coherence Scale (SOC) measure overall health and experience of context. Depression and anxiety are measured with Hospital Anxiety Depression Scale (HADS), schizotypic traits with SPQ and obsessive symptoms are assessed with BOCS. Suicide thoughts are examined using one item in PHQ-9 in addition to structured questions about suicidal thoughts included in the structured diagnostic interview material M.I.N.I. (version 7.0.0). The self-assessment form RAADS - Ritvo Autism-Asperger's Diagnostic Scale is used to measure autistic traits. Knowledge about autism is measured before, during and after treatment using Autism Knowledge questionnaire, which is a questionnaire created for the project. Self-acceptance, self-awareness, mood and ability to ask for help, as well as the extent of social contacts, sickness absence, and occurrence of work / studies will be measured before and after the intervention using a battery of questions compiled for the project. Satisfaction with the treatment is measured with CSQ and negative side effects are measured through Negative Effects questionnaire (NEQ) after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have ASD diagnosis
* Must have normal IQ
* Must be able to understand and read swedish

Exclusion Criteria:

* high risk of suicide
* psychosis
* inability to fill out forms and answer questions on the internet
* inability to read and understand the Swedish language
* ongoing psychotherapy with CBT or social behavior training
* mental development disorder

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Change in life quality | Change from Baseline, at 9 weeks, at 18 weeks, at 6 months and at 12 months
  Possible interaction effect between group and time in respect of differences in quality of life of the intervention group and the control group between pre, post and follow-up measurement
Change in Sense of coherence | Change from Baseline, at 18 weeks, at 6 months and at 12 months
  Possible interaction effect between group and time in respect of differences in Sense of coherence of the intervention group and the control group between pre, post and follow-up measurement. Sense of coherence will be measured using SOC-13 questionnaire.

SECONDARY OUTCOMES:
Change in depressive and anxiety symptoms | Change from Baseline, at 9 weeks, at 18 weeks, at 6 months and at 12 months
  Possible interaction effect between group and time in respect of differences in Depressive and anxiety symptoms of the intervention group and the control group between pre, post and follow-up measurement. Depression and anxiety symptoms will be measured using HADS
Subjective experience of ICBT | At 19 weeks
  The subjective experience of participating in an internet based treatment will be qualitatively evaluated using semi structured interview.
Content of communication | At 20 weeks
  Thematic content of the written communication between participant and therapist will be assessed using content analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Britta Westerberg, Principal Investigator — Region Örebro County
Locations (1):
- Region Örebro County, Örebro, Örebro County, Sweden

REFERENCES:
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Ware, JE., Kosinski, M. & Gandek, B. (2005). SF-36 health survey: Manual and interpretation guide. Lincoln: Quality Metric, Inc.
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Shulte, D., (2005). Zeitschrift für Klinische Psychologie und Psychotherapie, 34, 176-188.
- [Background] Sheehan, D.V., Lecrubier, Y., Sheehan, K., Harnett, J., Weiller, E., Keskiner, A., Schinka, J., Knapp, E., Sheehan, M. F. & Dunbar, G. C. (1997). Reliability and validity of the Mini International Neuropsychiatric Interview (M.I.N.I.) according to the SCID-P. European Psychiatry, Vol 12(5), 1997, 232-241
- [Background] Rydén, E. & Bejerot, S. (2008). Autism Spectrum Disorders in an adult Psychiatric Population. A Naturalistic Cross-Sectional controlled study. Clinical Neuropsychiatry, 5, 1, 13-21.
- [Background] Rozental A, Kottorp A, Boettcher J, Andersson G, Carlbring P. Negative Effects of Psychological Treatments: An Exploratory Factor Analysis of the Negative Effects Questionnaire for Monitoring and Reporting Adverse and Unwanted Events. PLoS One. 2016 Jun 22;11(6):e0157503. doi: 10.1371/journal.pone.0157503. eCollection 2016. PMID 27331907
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Ramsay, JR., Brodkin, R. Cohen, ES. Listerud, MR. & Rostain, J. (2005). "Better Strangers": Using the Relationship in Psychotherapy for Adult Patients with Asperger Syndrome. Psychotherpy: Theory, Research, Practice, Training, 42, 483-93
- [Background] Raine, A., & Benishay, D (1995). The SPQ-B: A Brief Screening Instrument for Schizotypal Personality Disorder. Journal of Personality Disorders: Vol. 9, No. 4, pp. 346-355.
- [Background] Martin PJ, Sterne AL. Prognostic expectations and treatment outcome. J Consult Clin Psychol. 1975 Aug;43(4):572-6. doi: 10.1037/h0076886. No abstract available. PMID 1159154
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Howlin, P. (2003). Autism preparing for adulthood. London: Routledge.
- [Background] Howlin, P. (2000). Outcome in adult life for more able individuals with autism or Asperger syndrome. Autism, 4, 63-83
- [Background] Hesselmark E, Plenty S, Bejerot S. Group cognitive behavioural therapy and group recreational activity for adults with autism spectrum disorders: a preliminary randomized controlled trial. Autism. 2014 Aug;18(6):672-83. doi: 10.1177/1362361313493681. Epub 2013 Oct 2. PMID 24089423
- [Background] Guy, W. (1976). The Clinical Global Impression Scale. ECDEU Assessment Manual for Psychopharmacology. 218-222
- [Background] Gaus, LV. (2007). Cognitive-Behavioral Therapy for Adult Asperger Syndrome. New York, NY: Guilford Press.
- [Background] Frith U, Happe F. Autism: beyond "theory of mind". Cognition. 1994 Apr-Jun;50(1-3):115-32. doi: 10.1016/0010-0277(94)90024-8. PMID 8039356
- [Background] Frisch, MB., Cornell, Villanueva & Retzlaff. (1992). Clinical validation of the Quality of Life Inventory. A measure of life satisfaction for use in treatment planning and outcome assessment. Psychol Assess, 4, 92-101.
- [Background] Bejerot S, Eriksson JM, Mortberg E. Social anxiety in adult autism spectrum disorder. Psychiatry Res. 2014 Dec 15;220(1-2):705-7. doi: 10.1016/j.psychres.2014.08.030. Epub 2014 Aug 27. PMID 25200187
- [Background] Bejerot S, Edman G, Anckarsater H, Berglund G, Gillberg C, Hofvander B, Humble MB, Mortberg E, Rastam M, Stahlberg O, Frisen L. The Brief Obsessive-Compulsive Scale (BOCS): a self-report scale for OCD and obsessive-compulsive related disorders. Nord J Psychiatry. 2014 Nov;68(8):549-59. doi: 10.3109/08039488.2014.884631. Epub 2014 Feb 25. PMID 24568661
- [Background] Attwood T. (2008). Den kompletta guiden till Aspergers syndrom. Stockholm: Cura.
- [Background] Antonovsky A. The structure and properties of the sense of coherence scale. Soc Sci Med. 1993 Mar;36(6):725-33. doi: 10.1016/0277-9536(93)90033-z. PMID 8480217
- [Background] Andersen LM, Naswall K, Manouilenko I, Nylander L, Edgar J, Ritvo RA, Ritvo E, Bejerot S. The Swedish version of the Ritvo autism and asperger diagnostic scale: revised (RAADS-R). A validation study of a rating scale for adults. J Autism Dev Disord. 2011 Dec;41(12):1635-45. doi: 10.1007/s10803-011-1191-3. PMID 21327833
- [Derived] Westerberg B, Jacobson K, Unenge Hallerback M, Bejerot S, Hollandare F. Communicative Behaviors in an Internet-Based Intervention for Individuals With Autism: Mixed Methods Analysis. J Med Internet Res. 2026 Feb 4;28:e76527. doi: 10.2196/76527. PMID 41637734
- [Derived] Klang A, Westerberg B, Humble MB, Bejerot S. The impact of schizotypy on quality of life among adults with autism spectrum disorder. BMC Psychiatry. 2022 Mar 19;22(1):205. doi: 10.1186/s12888-022-03841-2. PMID 35305592